CLINICAL TRIAL: NCT02664142
Title: Monitoring the Depth of Anaesthesia in Children in the Course of a Surgical Procedure Using the BIS Monitor - Prospective Randomized Study
Brief Title: BIS Monitoring of the Depth of Anaesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNO-KARIM-3
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: General Surgery; Anaesthesia
Keywords: General Surgery; Child; Anaesthesia; Depth of anaesthesia; BIS monitoring
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS Group (Experimental): BIS monitor will be used during the GA monitoring, the BIS value will be known to the anaesthetist (investigator)
  * GA induction (Phase 1):
    1. inhalation introduction (Sevorane, 02,AIR (flow 2:2 l/min)) or
    2. intra-venous introduction: (Suphentanil: (0.1-0.3 ug/kg iv.), Propofol (2-2,5 mg/kg iv.), or Mivacron (0.15-2mg/kg ),Tracrium (0.3-0.6mg/kg)
  * anaesthesia (Phase 2, Phase 3):
    1. hypnotic component: titration of Sevorane concentration, with the aim of achieving the BIS values of 40-60%, bearing gas mixture: O2/AIR (in proportion of 1:1, with 0.5:0.5 flows)
    2. analgesic component: Suphentanil (continuous dose of 0.1-0.3ug/kg iv. every 20-30 min)
    3. relaxation: Mivacron (continuous dose of 0.1mg/kg iv.), Tracrium(0.3-0.6 mg/kg) Patients in this group will be administered anaesthetic, in order to achieve and maintain the required general anaesthesia.
  Interventions: Procedure: BIS Group; Drug: Anaesthetics
- Non-BIS Group (Experimental): BIS monitor will be used during the GA monitoring, however the BIS value will not be known to the anaesthetist (investigator)
  * GA induction (Phase 1):
    1. inhalation introduction (Sevorane, 02,AIR (flow 2:2 l/min)) or
    2. intra-venous introduction: (Suphentanil: (0.1-0.3 ug/kg iv.), Propofol (2-2,5 mg/kg iv.), or Mivacron (0.15-2mg/kg ),Tracrium (0.3-0.6mg/kg)
  * anaesthesia (Phase 2, Phase 3):
    1. hypnotic component: titration of Sevorane concentration, with the aim of achieving the MAC value appropriate for the age of the child, bearing gas mixture: O2/AIR (in proportion of 1:1, with 0.5:0.5 flows)
    2. analgesic component: Suphentanil (continuous dose of 0.1-0.3ug/kg iv. every 20-30 min)
    3. relaxation: Mivacron (continuous dose of 0.1mg/kg iv.), Tracrium(0.3-0.6 mg/kg) Patients in this group will be administered anaesthetic, in order to achieve and maintain the required general anaesthesia.
  Interventions: Procedure: Non-BIS Group; Drug: Anaesthetics

INTERVENTIONS:
Procedure: BIS Group — BIS monitoring will be used in the BIS Group patients. The BIS value will be known to the anaesthetist, who will be able to act accordingly.
  Arms: BIS Group
Procedure: Non-BIS Group — BIS monitoring will be used in the Non-BIS Group patients. The BIS value will NOT be known to the anaesthetist and will be observed by a trained co-investigator, with subsequent evaluation.
  Arms: Non-BIS Group
Drug: Anaesthetics — Anaesthetics will be administered in both experimental groups, in order to maintain the required general anaesthesia.

SUMMARY:
General anaesthesia (GA) is, according to many definitions, the greatest gift presented to the medical art (S. B. Nuland). One of the aims of GA is to achieve the optimal depth of anaesthesia and rapid emergence from general anaesthesia. In order to achieve this goal, it is necessary to observe the clinical condition of the patient, and at the same time monitor the patient's overall condition. With the currently available options of GA management (e.g. use of intravenous anaesthetics, strong analgesics and modern volatile anaesthetics, in combination with various methods of topical anaesthesia) the importance of methods measuring the depth of GA increases. The depth of GA may be defined as a continuous progressive decreasing of the central nervous system, together with a decreased reactivity to stimuli. In the course of GA, perioperative awareness is detected in 0.1-0.2% of cases. Awakening during a surgical procedure may result in significant psychological complications (e.g. post-traumatic stress disorder), and the patient may suffer from a serious long-time disorder.

DETAILED DESCRIPTION:
In order to prevent, or minimize the perioperative awareness, it is possible to utilize two different methods of depth of anaesthesia monitoring. The options may be divided into two basic groups: A/ The use of clinical monitoring and other methods (apart from CNS), and B/ Methods based on monitoring of the electrical activity of the brain. In the first group, it is possible to list the following options: 1. clinical assessment (Evans's score), 2. skin conductance, 3. isolated method of measurement at the forearm, 4. spontaneous superficial electromyogram (SEMG), 5. lower oesophageal contractility, and 6. various hearth rate. The possibilities of depth of GA monitoring using the scanning of electrical brain activity may be further subdivided into two groups: a/ methods based on EEG, and b/ methods assessing evoked potentials. In the group of methods based on EEG, the following devices may be used to monitor the depth of GA in practice:

a/ BIS monitor, b/ E-Entropy, c/ Narcotrend, and d/ SedLine Sedation Monitor. In the second group using evoked potentials it is possible to utilize monitors measuring electrical activity in certain areas of the brain, in relation to stimulation of specific sensory nerve pathways: a/ somatosensory, b/ visual, and c/ auditive evoked potentials.

Aims of the Study:

Null hypothesis: The use of depth of general anaesthesia monitoring in children in the course of a surgical procedure does not affect the number of post-operative complications related to the depth of GA, does not shorten the period of emergence from GA, does not decrease the amount of inhalation anaesthetics used, and does not decrease the amount of opioids used.

Primary aim: To test, whether the administration of anaesthesia in children in the course of a surgical procedure with the depth of general anaesthesia monitoring with the BIS monitor results in a decrease in the number of complications related to inappropriate depth of GA.

Secondary aim: To verify, whether the administration of anaesthesia in children in the course of a surgical procedure with the depth of general anaesthesia monitoring with the BIS monitor:

1. results in a shortening of the emergence from general anaesthesia
2. results in a decrease in the amount of inhalation anaesthetic used
3. results in a decrease in the amount of analgesics used

Tertiary aim: To verify, whether the administration of general anaesthesia in children in the course of a surgical procedure with the depth of general anaesthesia monitoring with the BIS monitor:

a/results in a decrease of early post-operative complications at the recovery room.

Study design:

Procedure to achieve the study aims The study is a prospective, interventional study, performed at the Anaesthesiology-Resuscitation Department of the University Hospital Ostrava. The study has been approved by the Head of the Department, prof. Pavel Ševčík, MD, CSc. Furthermore, the study has been approved by the Ethics Committee of the University Hospital Ostrava and is in compliance with the principles of the Declaration of Helsinki. Informed consent will be obtained for every paediatric patient, the Informed consent form has also been approved by the Ethics Committee, and will be signed by both parents.

The study group will include paediatric patients at the age from 28 days to 15 years of age (including), ASA I classification.

Interventional arm of the study will be characterized by the BIS monitoring and management of the hypnotic component of general anaesthesia towards the values of BIS 40-60.

Conventional arm of the study will be performed without the depth of anaesthesia monitoring (however, the BIS value will be recorded by an independent participant), and management of the hypnotic component of general anaesthesia according to MAC value appropriate for the age of the child.

Each study arm will include the total of 100 paediatric study subjects. Randomization will be performed by the envelope method.

Definition of terms

* BIS group: group of patients, in whom the hypnotic component of GA will be managed towards the value of BIS 40-60.
* Non-BIS group: group of patients, in whom the hypnotic component of GA will be managed towards the MAC value appropriate for the age of the child. Depth of GA will be also monitored with the BIS monitor, however, the BIS value will be unknown to the investigator.
* Period of emergence from anaesthesia: time interval from the moment of setting the zero concentration of inhalation anaesthetics on the vaporizer to the moment when the child manifests the signs of complete awareness: spontaneous ventilation, spontaneous motility, rising of the head, clasping of the hand, or crying.
* Consumption of inhalation anaesthetic: consumption of inhalation anaesthetic will be measured in two follow-up time phases of GA:

  1. Phase 1: from the moment when administration of the inhalation anaesthetic is initiated to the moment when breathing passageways are secured (LM, OTI). This phase of GA is characterized with a higher concentration of the inhalation anaesthetic and standard flows: O2, AIR in proportion of 2:2 l/min,
  2. Phase 2: continues after Phase 1, from the moment when breathing passageways are secured to the moment, when the zero value is set on the vaporizer. This phase of GA is characterized with gas flows: O2, AIR in proportion of 0.5:0.5 l/min.
* Consumption of analgesics: the amount of analgesics used during GA
* Early post-operative complications (assessed in the recovery room): the need of re-intubation, need to apply antidotes, laryngospasm, bronchospasm, hyperalgesia (pain assessment according to standard scales), vomiting
* Emergence from GA (Phase 3): continues after Phase 2, from the moment when the zero value is set on the vaporizer to the moment of LM or intubation cannula removal.

5.2.2. Protocol of GA management in the "BIS group": BIS monitor will be used during the GA monitoring, the BIS value will be known to the anaesthetist (investigator)

* GA induction (Phase 1):

  1. inhalation introduction (Sevorane, 02,AIR (flow 2:2 l/min)) or
  2. intra-venous introduction: (Suphentanil: (0.1-0.3 ug/kg iv.), Propofol (2-2,5 mg/kg iv.), or Mivacron (0.15-2mg/kg ),Tracrium (0.3-0.6mg/kg)
* anaesthesia (Phase 2, Phase 3):

  1. hypnotic component: titration of Sevorane concentration, with the aim of achieving the BIS values of 40-60%, bearing gas mixture: O2/AIR (in proportion of 1:1, with 0.5:0.5 flows)
  2. analgesic component: Suphentanil (continuous dose of 0.1-0.3ug/kg iv. every 20-30 min)
  3. relaxation: Mivacron (continuous dose of 0.1mg/kg iv.), Tracrium(0.3-0.6 mg/kg) 5.2.3. Protocol of GA management in the "Non-BIS group" BIS monitor will be used during the GA monitoring, however the BIS value will not be known to the anaesthetist (investigator)
* GA induction (Phase 1):

  1. inhalation introduction (Sevorane, 02,AIR (flow 2:2 l/min)) or
  2. intra-venous introduction: (Suphentanil: (0.1-0.3 ug/kg iv.), Propofol (2-2,5 mg/kg iv.), or Mivacron (0.15-2mg/kg ),Tracrium (0.3-0.6mg/kg)
* anaesthesia (Phase 2, Phase 3):

  1. hypnotic component: titration of Sevorane concentration, with the aim of achieving the MAC value appropriate for the age of the child, bearing gas mixture: O2/AIR (in proportion of 1:1, with 0.5:0.5 flows)
  2. analgesic component: Suphentanil (continuous dose of 0.1-0.3ug/kg iv. every 20-30 min)
  3. relaxation: Mivacron (continuous dose of 0.1mg/kg iv.), Tracrium(0.3-0.6 mg/kg)

Assessment:

The following parameters will be observed in the "BIS group" and the "Non-BIS group":

* occurrence of perioperative complications
* period of emergence from GA
* consumption of opioids
* consumption of inhalation anaesthetic
* occurrence of early post-operative complications at the recovery room
* BIS value

Statistical processing:

The obtained statistical data will be processed using statistical methods and presented in the form of tables and charts.

ELIGIBILITY:
Inclusion Criteria:

* appropriate age
* informed consent form signed by both parents (according to national legislation)
* need to undergo a procedure in general anaesthesia
* ASA I classification

Exclusion Criteria:

* non-signing of the informed consent form by both parents
* ASA classification higher than I

Ages: 15 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of perioperative complications | 24 months
  The occurrence of perioperative complications due to inappropriate depth of general anaesthesia will be observed.

SECONDARY OUTCOMES:
Shortening of the emergence from general anaesthesia | 24 months
  The time of emergence from general anaesthesia will be measured and compared in both groups.
Decrease in the amount of inhalation anaesthetic used | 24 months
  The decrease in the amount of inhalation anaesthetic used will be measured and compared in both groups.
Decrease in the amount of analgesics used | 24 months
  The decrease in the amount of analgesics used will be measured and compared in both groups.

OTHER OUTCOMES:
Decrease of complications at recovery room | 24 months
  The decrease in complications at recovery room will be measured and compared in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Divak, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No